CLINICAL TRIAL: NCT02060188
Title: A Phase 2 Clinical Trial of Nivolumab, or Nivolumab Combinations in Recurrent and Metastatic Microsatellite Instability High (MSI-H) and Non-MSI-H Colon Cancer
Brief Title: A Study of Nivolumab Alone or Nivolumab Combination Therapy in Colon Cancer That Has Come Back or Has Spread
Acronym: CheckMate142
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-142; 2013-003939-30 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2014-02-11 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Microsatellite Unstable Colorectal Cancer; Microsatellite Stable Colorectal Cancer; Mismatch Repair Proficient Colorectal Cancer; Mismatch Repair Deficient Colorectal Cancer
MeSH Terms: interventions — Ipilimumab; Nivolumab; cobimetinib; daratumumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Nivolumab Monotherapy (Experimental)
  Interventions: Drug: Nivolumab
- Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Nivolumab + Ipilimumab Cohort C3 (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Nivolumab + Ipilimumab + Cobimetinib Cohort C4 (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Cobimetinib
- Nivolumab + BMS-986016 Cohort C5 (Experimental)
  Interventions: Drug: Nivolumab; Drug: BMS-986016
- Nivolumab + Daratumumab Cohort C6 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Daratumumab

INTERVENTIONS:
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Nivolumab + Ipilimumab; Nivolumab + Ipilimumab + Cobimetinib Cohort C4; Nivolumab + Ipilimumab Cohort C3
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Drug: Cobimetinib — Specified dose on specified days
  Other Names: Cotellic
  Arms: Nivolumab + Ipilimumab + Cobimetinib Cohort C4
Drug: Daratumumab — Specified dose on specified days
  Other Names: Darzalex
  Arms: Nivolumab + Daratumumab Cohort C6
Drug: BMS-986016 — Specified dose on specified days
  Arms: Nivolumab + BMS-986016 Cohort C5

SUMMARY:
The purpose of this study is to examine if Nivolumab by itself, or Nivolumab in combination with other anti-cancer drugs, will result in meaningful tumor size reduction, in participants with colon cancer that has come back or has spread, and who have a specific biomarker in their tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Histologically confirmed recurrent or metastatic colorectal cancer
* Measurable disease per RECIST v1.1
* Microsatellite instability expression detected by an accredited laboratory
* Participants enrolled into the C3 Cohort must have not had treatment for their metastatic disease

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases are not allowed
* Prior treatment with an anti-Programmed Death Receptor (PD)-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-Cell Lymphoma-4 Antigen (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Prior malignancy active within the previous 3 years except for locally curable cancers
* Participants with active, known or suspected autoimmune disease
* Participants with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (14):
  - Local Institution - 0028, Gilbert, Arizona
  - Local Institution - 0004, Los Angeles, California
  - Local Institution - 0001, San Francisco, California
  - Local Institution - 0008, Atlanta, Georgia
  - Local Institution - 0002, Boston, Massachusetts
  - Local Institution - 0036, Boston, Massachusetts
  - Local Institution - 0034, Minneapolis, Minnesota
  - Local Institution - 0024, Durham, North Carolina
  - Local Institution - 0029, Winston-Salem, North Carolina
  - Local Institution - 0005, Portland, Oregon
  - Local Institution - 0041, Allentown, Pennsylvania
  - Local Institution - 0013, Pittsburgh, Pennsylvania
  - Local Institution - 0006, Nashville, Tennessee
  - Local Institution - 0003, Houston, Texas
- Australia (3):
  - Local Institution - 0040, Westmead, New South Wales
  - Local Institution - 0039, Southport, Queensland
  - Local Institution - 0037, Melbourne, Victoria
- Belgium (3):
  - Local Institution - 0019, Brussels
  - Local Institution - 0018, Brussels
  - Local Institution - 0020, Leuven
- Canada (2):
  - Local Institution - 0027, Edmonton, Alberta
  - Local Institution - 0016, Toronto, Ontario
- Local Institution - 0025, Paris, France
- Ireland (3):
  - Local Institution - 0022, Dublin
  - Local Institution - 0023, Dublin
  - Local Institution - 0033, Galway
- Italy (3):
  - Local Institution - 0030, Candiolo, Torino
  - Local Institution - 0035, Modena
  - Local Institution - 0032, Padua
- Spain (3):
  - Local Institution - 0012, Madrid, Madrid
  - Local Institution - 0010, Madrid
  - Local Institution - 0011, Seville

REFERENCES:
- [Derived] Overman MJ, Gelsomino F, Aglietta M, Wong M, Limon Miron ML, Leonard G, Garcia-Alfonso P, Hill AG, Cubillo Gracian A, Van Cutsem E, El-Rayes B, McCraith SM, He B, Lei M, Lonardi S. Nivolumab plus relatlimab in patients with previously treated microsatellite instability-high/mismatch repair-deficient metastatic colorectal cancer: the phase II CheckMate 142 study. J Immunother Cancer. 2024 May 31;12(5):e008689. doi: 10.1136/jitc-2023-008689. PMID 38821718
- [Derived] Lenz HJ, Van Cutsem E, Luisa Limon M, Wong KYM, Hendlisz A, Aglietta M, Garcia-Alfonso P, Neyns B, Luppi G, Cardin DB, Dragovich T, Shah U, Abdullaev S, Gricar J, Ledeine JM, Overman MJ, Lonardi S. First-Line Nivolumab Plus Low-Dose Ipilimumab for Microsatellite Instability-High/Mismatch Repair-Deficient Metastatic Colorectal Cancer: The Phase II CheckMate 142 Study. J Clin Oncol. 2022 Jan 10;40(2):161-170. doi: 10.1200/JCO.21.01015. Epub 2021 Oct 12. PMID 34637336
- [Derived] Overman MJ, Lonardi S, Wong KYM, Lenz HJ, Gelsomino F, Aglietta M, Morse MA, Van Cutsem E, McDermott R, Hill A, Sawyer MB, Hendlisz A, Neyns B, Svrcek M, Moss RA, Ledeine JM, Cao ZA, Kamble S, Kopetz S, Andre T. Durable Clinical Benefit With Nivolumab Plus Ipilimumab in DNA Mismatch Repair-Deficient/Microsatellite Instability-High Metastatic Colorectal Cancer. J Clin Oncol. 2018 Mar 10;36(8):773-779. doi: 10.1200/JCO.2017.76.9901. Epub 2018 Jan 20. PMID 29355075
- [Derived] Overman MJ, McDermott R, Leach JL, Lonardi S, Lenz HJ, Morse MA, Desai J, Hill A, Axelson M, Moss RA, Goldberg MV, Cao ZA, Ledeine JM, Maglinte GA, Kopetz S, Andre T. Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. Lancet Oncol. 2017 Sep;18(9):1182-1191. doi: 10.1016/S1470-2045(17)30422-9. Epub 2017 Jul 19. PMID 28734759
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Nivolumab Monotherapy: Nivolumab 3 mg/kg
- Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg
- Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg twice in six weeks Q6W
- MSS: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W
- Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
- Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg
- Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg
- Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg: Nivolumab 240 mg + BMS-986016 80 mg
- Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg: Nivolumab FD + Daratumumab 16 mg/kg
Period: Overall Study
Arm/Group | Cohort 1: Nivolumab Monotherapy | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | MSS: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg
Started | 74 | 119 | 45 | 10 | 10 | 3 | 30 | 50 | 44
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 74 | 119 | 45 | 10 | 10 | 3 | 30 | 50 | 44
Not completed — Disease Progression | 36 | 42 | 8 | 5 | 6 | 3 | 23 | 20 | 43
Not completed — Study Drug Toxicity | 10 | 18 | 7 | 4 | 3 | 0 | 2 | 5 | 0
Not completed — Adverse event unrelated to study drug | 2 | 5 | 6 | 0 | 1 | 0 | 4 | 4 | 1
Not completed — Participant request to discontinue study treatment | 7 | 7 | 4 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Participant withdrew consent | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 13 | 38 | 19 | 0 | 0 | 0 | 0 | 10 | 0
Not completed — Other reason | 3 | 7 | 0 | 1 | 0 | 0 | 0 | 9 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Administrative reasons by sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nivolumab Monotherapy | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | MSS: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg | Total
Number analyzed (Participants) | 74 | 119 | 45 | 10 | 10 | 3 | 30 | 50 | 44 | 385
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 57 | 81 | 22 | 9 | 9 | 3 | 21 | 34 | 32 | 268
  >= 65 and < 75 years | 13 | 27 | 10 | 1 | 1 | 0 | 9 | 10 | 9 | 80
  >= 75 years | 4 | 11 | 13 | 0 | 0 | 0 | 0 | 6 | 3 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 49 | 22 | 2 | 3 | 1 | 12 | 22 | 14 | 155
  Male | 44 | 70 | 23 | 8 | 7 | 2 | 18 | 28 | 30 | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 110 | 43 | 10 | 10 | 3 | 23 | 49 | 41 | 354
  Black or African American | 7 | 2 | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 16
  Asian | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 7
  Other | 1 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 7
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Per Investigator Assessment
Description: Objective Response Rate (ORR) is defined as the number of randomized participants who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on investigator assessments [using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1], divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization to the date of objectively documented progression or the date of subsequent systemic cancer therapy, whichever occurs first (Up to approximately 127 months)
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg: Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg
Arm/Group | Cohort 1: Nivolumab Monotherapy | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg | MSS: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 74 | 119 | 45 | 30 | 50 | 44 | 10 | 3 | 10
percentage of participants | 40.5 [29.3 to 52.6] | 66.4 [57.2 to 74.8] | 71.1 [55.7 to 83.6] | 3.3 [0.1 to 17.2] | 50.0 [35.5 to 64.5] | 0 [0.0 to 8.0] | 0 [0.0 to 25.9] | 0 [0.0 to 63.2] | 10.0 [0.5 to 39.4]

2. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Per Independent Review Committee (IRC)
Description: Objective Response Rate (ORR) is defined as the number of randomized participants who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on IRC[using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1], divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: All treated participants. As pre-specified only applicable for Cohort 1, 2, 3, 4, 5 and 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab Monotherapy | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg
Number analyzed (Participants) | 74 | 119 | 45 | 30 | 50 | 44
percentage of participants | 37.8 [26.8 to 49.9] | 61.3 [52.0 to 70.1] | 62.2 [46.5 to 76.2] | 6.7 [0.8 to 22.1] | 50.0 [35.5 to 64.5] | 0 [0.0 to 8.0]

ADVERSE EVENTS:
Time Frame: From Day 1 and up to approximately 127 months.
Description: All treated participants
Groups:
- MSS Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: MSS: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W
- Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg: Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg
Arm/Group | Cohort 1: Nivolumab Monotherapy | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W | MSS Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg
All-Cause Mortality (participants affected / at risk) | 44/74 | 46/119 | 16/45 | 9/10 | 3/3 | 10/10 | 29/30 | 27/50 | 43/44
Serious Adverse Events (participants affected / at risk) | 46/74 | 72/119 | 22/45 | 8/10 | 3/3 | 9/10 | 20/30 | 28/50 | 29/44
Other Adverse Events (participants affected / at risk) | 73/74 | 116/119 | 45/45 | 10/10 | 3/3 | 10/10 | 27/30 | 48/50 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nivolumab Monotherapy (N=74) | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=119) | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W (N=45) | MSS Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=10) | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg (N=3) | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=10) | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg (N=30) | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg (N=50) | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular myasthenia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 3 | 3 | 0 | 0 | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders and administration site conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders and administration site conditions) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Incarcerated hernia (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders and administration site conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain (General disorders and administration site conditions) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders and administration site conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders and administration site conditions) | 2 | 4 | 4 | 1 | 0 | 1 | 1 | 0 | 2
Stenosis (General disorders and administration site conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders and administration site conditions) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Suprapubic pain (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis infective (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metapneumovirus pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Pseudomonas infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal deviation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 12 | 3 | 5 | 2 | 2 | 9 | 9 | 19
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis in device (Product issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nivolumab Monotherapy (N=74) | Cohort 2: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=119) | Cohort 3: Nivolumab 3 mg/kg Q2W with Ipilimumab 1 mg/kg Q6W (N=45) | MSS Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (N=10) | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg (N=3) | Non-MSI-H: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=10) | Cohort 4: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg + Cobimetinib 60 mg (N=30) | Cohort 5: Nivolumab 240 mg + BMS-986016 80 mg (N=50) | Cohort 6: Nivolumab FD + Daratumumab 16 mg/kg (N=44)
Anaemia (Blood and lymphatic system disorders) | 33 | 41 | 10 | 1 | 0 | 4 | 14 | 9 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 9 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 16 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 5 | 5 | 1 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 8 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 4 | 18 | 6 | 0 | 0 | 0 | 1 | 2 | 0
Hypothyroidism (Endocrine disorders) | 9 | 22 | 10 | 0 | 0 | 0 | 3 | 8 | 2
Dry eye (Eye disorders) | 2 | 5 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Serous retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 5 | 5 | 3 | 1 | 0 | 1 | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 6 | 1 | 1 | 1 | 1 | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 28 | 37 | 14 | 2 | 0 | 3 | 2 | 7 | 12
Abdominal pain lower (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 12 | 16 | 5 | 1 | 0 | 1 | 2 | 6 | 5
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 20 | 27 | 7 | 2 | 0 | 2 | 4 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 43 | 73 | 20 | 4 | 0 | 4 | 19 | 18 | 18
Dry mouth (Gastrointestinal disorders) | 4 | 11 | 5 | 2 | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 11 | 7 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 3 | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 5 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 36 | 39 | 17 | 3 | 1 | 4 | 10 | 9 | 15
Stomatitis (Gastrointestinal disorders) | 6 | 6 | 4 | 0 | 0 | 0 | 2 | 6 | 0
Toothache (Gastrointestinal disorders) | 3 | 11 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 30 | 31 | 14 | 4 | 0 | 4 | 7 | 9 | 6
Asthenia (General disorders and administration site conditions) | 18 | 38 | 14 | 2 | 0 | 3 | 0 | 18 | 11
Chills (General disorders and administration site conditions) | 5 | 9 | 2 | 0 | 0 | 2 | 3 | 1 | 4
Fatigue (General disorders and administration site conditions) | 39 | 43 | 15 | 5 | 2 | 5 | 13 | 5 | 10
Feeling of body temperature change (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders and administration site conditions) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Influenza like illness (General disorders and administration site conditions) | 3 | 17 | 2 | 0 | 0 | 0 | 1 | 6 | 5
Mucosal inflammation (General disorders and administration site conditions) | 2 | 6 | 3 | 1 | 0 | 1 | 1 | 1 | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 9 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders and administration site conditions) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders and administration site conditions) | 13 | 13 | 5 | 1 | 1 | 1 | 6 | 2 | 4
Pain (General disorders and administration site conditions) | 4 | 14 | 6 | 2 | 0 | 0 | 1 | 4 | 0
Pyrexia (General disorders and administration site conditions) | 25 | 52 | 15 | 2 | 0 | 5 | 4 | 18 | 13
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 5
Eye infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 7 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 10 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 14 | 21 | 7 | 0 | 0 | 0 | 0 | 5 | 2
Oral candidiasis (Infections and infestations) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 12 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 14 | 3 | 0 | 0 | 0 | 0 | 3 | 3
Urinary tract infection (Infections and infestations) | 10 | 14 | 3 | 0 | 0 | 0 | 4 | 2 | 1
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 10 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 3 | 1 | 0 | 0 | 1 | 5 | 17
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 13 | 24 | 7 | 1 | 1 | 2 | 8 | 1 | 3
Amylase increased (Investigations) | 10 | 19 | 7 | 0 | 0 | 0 | 2 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 13 | 28 | 4 | 1 | 1 | 2 | 12 | 1 | 2
Blood albumin decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 10 | 10 | 3 | 0 | 1 | 1 | 15 | 0 | 4
Blood bilirubin increased (Investigations) | 7 | 7 | 2 | 0 | 2 | 1 | 5 | 2 | 5
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 1 | 0 | 0 | 0 | 15 | 1 | 0
Blood creatinine increased (Investigations) | 6 | 20 | 9 | 0 | 0 | 0 | 3 | 7 | 2
Blood magnesium decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood potassium increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 3 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Blood sodium increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 14 | 24 | 8 | 0 | 0 | 0 | 6 | 5 | 1
Lymphocyte count decreased (Investigations) | 4 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Platelet count decreased (Investigations) | 6 | 6 | 2 | 0 | 0 | 0 | 8 | 1 | 0
Transaminases increased (Investigations) | 0 | 5 | 2 | 0 | 0 | 1 | 0 | 2 | 1
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Weight decreased (Investigations) | 8 | 14 | 7 | 0 | 1 | 3 | 3 | 4 | 3
Weight increased (Investigations) | 9 | 10 | 3 | 0 | 0 | 0 | 0 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 31 | 11 | 4 | 1 | 7 | 10 | 14 | 11
Dehydration (Metabolism and nutrition disorders) | 7 | 9 | 3 | 1 | 0 | 3 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 9 | 3 | 1 | 1 | 1 | 1 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 9 | 8 | 0 | 0 | 1 | 0 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 1 | 1 | 1 | 9 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 6 | 1 | 0 | 1 | 0 | 2 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 11 | 2 | 0 | 1 | 2 | 8 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 11 | 3 | 1 | 0 | 1 | 7 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 9 | 1 | 2 | 0 | 3 | 3 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 31 | 16 | 2 | 0 | 0 | 1 | 15 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 36 | 8 | 1 | 1 | 2 | 2 | 5 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 7 | 3 | 0 | 0 | 0 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2 | 2 | 0 | 1 | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 13 | 5 | 0 | 0 | 0 | 3 | 6 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 9 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 14 | 10 | 1 | 0 | 2 | 1 | 3 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 11 | 13 | 5 | 1 | 1 | 1 | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 4 | 2 | 1 | 0 | 2 | 1 | 2 | 1
Headache (Nervous system disorders) | 17 | 25 | 5 | 2 | 0 | 1 | 4 | 4 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 9 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 7 | 10 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 9 | 14 | 5 | 0 | 0 | 1 | 0 | 2 | 3
Depressed mood (Psychiatric disorders) | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 6 | 4 | 0 | 0 | 1 | 1 | 3 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 26 | 9 | 4 | 1 | 1 | 1 | 6 | 1
Dysuria (Renal and urinary disorders) | 5 | 8 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Haematuria (Renal and urinary disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 43 | 10 | 3 | 2 | 2 | 7 | 8 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 20 | 7 | 5 | 2 | 4 | 6 | 5 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 1 | 0 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 4 | 0 | 1 | 0 | 4 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 3 | 0 | 0 | 0 | 1 | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 5 | 1 | 0 | 0 | 2 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 0 | 1 | 6 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 21 | 4 | 0 | 0 | 2 | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 11 | 2 | 1 | 0 | 0 | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 7 | 2 | 0 | 0 | 1 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 40 | 20 | 1 | 1 | 2 | 9 | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 16 | 26 | 12 | 1 | 1 | 2 | 8 | 6 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 10 | 3 | 0 | 0 | 0 | 6 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 5 | 3 | 0 | 0 | 1 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hot flush (Vascular disorders) | 6 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypertension (Vascular disorders) | 14 | 17 | 8 | 1 | 1 | 1 | 3 | 5 | 4
Hypotension (Vascular disorders) | 1 | 10 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 4 | 4 | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 7 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 6 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 5 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product issues) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT02060188/Prot_SAP_000.pdf